CLINICAL TRIAL: NCT04397237
Title: Prevalence, Seroconversion and Impact of COVID-19 in Autoimmune Diseases in Europe
Brief Title: Prevalence and Seroconversion of COVID-19 in Autoimmune Diseases in Europe
Acronym: Euro-COVIMID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pitié-Salpêtrière Hospital (Other)
Collaborators: Università degli Studi di Ferrara (Other); Rheumazentrum Ruhrgebiet (Other); University College, London (Other); University of Coimbra (Other); Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Pr David Saadoun, Principal Investigator, Pitié-Salpêtrière Hospital
Other Study IDs: 2020-A01371-38
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: COVID-19; Systemic Lupus Erythematosus; Sjogren's Syndrome; Axial Spondyloarthritis; Rheumatoid Arthritis; Giant Cell Arteritis
Keywords: COVID-19; Systemic Lupus Erythematosus; Sjogren's Syndrome; Axial Spondyloarthritis; Rheumatoid Arthritis; Giant Cell Arteritis; Prevalence
MeSH Terms: conditions — COVID-19; Lupus Erythematosus, Systemic; Sjogren's Syndrome; Axial Spondyloarthritis; Arthritis, Rheumatoid; Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Systemic Lupus Erythematosus: Consecutive Systemic Lupus Erythematosus patients followed-up in each service
- Sjogren's Syndrome: Consecutive Sjogren's Syndrome patients followed-up in each service
- Axial Spondyloarthritis: Consecutive Axial Spondyloarthritis patients followed-up in each service
- Rheumatoid Arthritis: Consecutive Rheumatoid Arthritis patients followed-up in each service
- Giant Cell Arteritis: Consecutive Giant Cell Arteritis patients followed-up in each service

SUMMARY:
The coronavirus disease 2019 (COVID-19) pandemic is a potentially fatal disease that represents a great global public health concern. In European countries such as Spain, Italy, Germany, Portugal, England and France, the pandemic has been of utmost importance. To date, no treatment has been robustly validated, and two theoretically opposite therapeutic strategies are proposed, based either on antiretroviral therapy or on immunomodulating agents.

In this complex context, people living with immune-mediated inflammatory diseases (IMID) raise specific concerns due to their potentially increased risk of infections or of severe infections. Among IMID, Sjögren's syndrome, systemic lupus erythematosus, rheumatoid arthritis, spondyloarthritis and giant cell arteritis are some key diseases.

In this cross-sectional, observational, multi-centric study, the investigators aim to assess both clinical and serological prevalence of COVID-19 among samples of IMID patients in Europe. In parallel, the investigators aim to compare the prevalence of COVID-19 seroconversion across these five IMIDs, their penetration across different 6 European countries (France, Italy, Spain, Germany, United Kingdom and Portugal), and to assess the severity of COVID-19 in these patients. Moreover, changes in treatment will be assessed, including immunomodulatory tapering or discontinuation, its causes over the outbreak period, as well as the incidence of IMID flares and their severity over this same period. Finally, patient's perceptions towards the pandemic will be evaluated and compared to medication beliefs.

Data will be collected through questionnaires during medical visit or phone consultation and serological tests will be performed within routine blood collection. As so, all study procedures are comprised within usual care. Through this study the investigators expect to have a better knowledge of the clinical and serological prevalence of COVID-19 in IMID across Europe, along with the psychological, clinical, and therapeutic impact of COVID-19 in this particular patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patients fitting classification criteria for each IMID (i.e., Sjögren's syndrome, systemic lupus erythematosus, rheumatoid arthritis, axial spondyloarthritis or giant cell arteritis);
* Willingness to participate;
* There are no specific inclusion criteria based on IMID previous activity, treatment or known COVID-19.

Exclusion Criteria:

* Patients who refuse to participate;
* Patients who don't speak or read the local language,
* Patients unable to perform a routine blood collection during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed-up for Sjögren's syndrome, systemic lupus erythematosus, rheumatoid arthritis, spondyloarthritis and giant cell arteritis in selected European tertiary-care centres will be contacted. The required number of patients with definite IMIDs who satisfy the inclusion criteria, followed-up in outpatient visits in the participating centres by one of the investigators, will be asked to participate. Consecutive patients fitting inclusion criteria will be selected in each centre in order to reduce bias selection.
Sampling Method: Non-Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
COVID-19 seroconversion | 1 day, during routine blood collection
  ELISA tests for COVID-19 antibodies
COVID-19 infection | During medical visit or phone consultation, up to 2 hours
  Case report form filled by the health professional

SECONDARY OUTCOMES:
Seroconversion rate by disease | 1 day, during routine blood collection
  Descriptive analysis for each disease's rate
Penetration across Europe | 1 day, during routine blood collection
  Descriptive analysis for each country's rate
COVID-19 severity | During medical visit, up to 1 hour
  World Health Organization ordinal scale for clinical improvement at any given point of the infection, going from 0 to 8, where higher scores means worse outcome.
COVID-19 mortality rate | During contact with family members, up to 1 hour
  Descriptive analysis for overall and COVID-19-linked mortality rates
COVID-19 impact on immunomodulatory treatment | During medical visit, up to 1 hour
  Case report form filled by the health professional
Patient-reported flares | During medical visit, up to 1 hour
  Case report form filled by the patient
Patient's fears towards COVID-19 | During medical visit, up to 1 hour
  Fear of COVID-19 scale, going from 7 to 35, where higher scores means worse outcome.
Patient's beliefs in their medicines towards COVID-19 | During medical visit, up to 1 hour
  Beliefs about Medicines Questionnaire, going from 11 to 55, with higher scores indicating stronger beliefs regarding medicine.

CONTACTS AND LOCATIONS:
Overall Officials: David Saadoun, MD, PhD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Saadoun, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pope JE. What Does the COVID-19 Pandemic Mean for Rheumatology Patients? Curr Treatm Opt Rheumatol. 2020;6(2):71-74. doi: 10.1007/s40674-020-00145-y. Epub 2020 Apr 30. PMID 32355607
- [Background] Favalli EG, Agape E, Caporali R. Incidence and Clinical Course of COVID-19 in Patients with Connective Tissue Diseases: A Descriptive Observational Analysis. J Rheumatol. 2020 Aug 1;47(8):1296. doi: 10.3899/jrheum.200507. Epub 2020 Apr 25. No abstract available. PMID 32335513
- [Background] Mathian A, Mahevas M, Rohmer J, Roumier M, Cohen-Aubart F, Amador-Borrero B, Barrelet A, Chauvet C, Chazal T, Delahousse M, Devaux M, Euvrard R, Fadlallah J, Florens N, Haroche J, Hie M, Juillard L, Lhote R, Maillet T, Richard-Colmant G, Palluy JB, Pha M, Perard L, Remy P, Riviere E, Sene D, Seve P, Morelot-Panzini C, Viallard JF, Virot JS, Benameur N, Zahr N, Yssel H, Godeau B, Amoura Z. Clinical course of coronavirus disease 2019 (COVID-19) in a series of 17 patients with systemic lupus erythematosus under long-term treatment with hydroxychloroquine. Ann Rheum Dis. 2020 Jun;79(6):837-839. doi: 10.1136/annrheumdis-2020-217566. Epub 2020 Apr 24. No abstract available. PMID 32332072
- [Background] Monti S, Balduzzi S, Delvino P, Bellis E, Quadrelli VS, Montecucco C. Clinical course of COVID-19 in a series of patients with chronic arthritis treated with immunosuppressive targeted therapies. Ann Rheum Dis. 2020 May;79(5):667-668. doi: 10.1136/annrheumdis-2020-217424. Epub 2020 Apr 2. No abstract available. PMID 32241793
- [Background] Gianfrancesco MA, Hyrich KL, Gossec L, Strangfeld A, Carmona L, Mateus EF, Sufka P, Grainger R, Wallace Z, Bhana S, Sirotich E, Liew J, Hausmann JS, Costello W, Robinson P, Machado PM, Yazdany J; COVID-19 Global Rheumatology Alliance Steering Committee. Rheumatic disease and COVID-19: initial data from the COVID-19 Global Rheumatology Alliance provider registries. Lancet Rheumatol. 2020 May;2(5):e250-e253. doi: 10.1016/S2665-9913(20)30095-3. Epub 2020 Apr 16. No abstract available. PMID 32309814
- [Background] Ahorsu DK, Lin CY, Imani V, Saffari M, Griffiths MD, Pakpour AH. The Fear of COVID-19 Scale: Development and Initial Validation. Int J Ment Health Addict. 2022;20(3):1537-1545. doi: 10.1007/s11469-020-00270-8. Epub 2020 Mar 27. PMID 32226353
- [Derived] Saadoun D, Vieira M, Vautier M, Baraliakos X, Andreica I, da Silva JAP, Sousa M, Luis M, Khmelinskii N, Gracia JMA, Castrejon I, Gonzalez JCN, Scire CA, Silvagni E, Bortoluzzi A, Penn H, Hamdulay S, Machado PM, Fautrel B, Cacoub P, Resche-Rigon M, Gossec L. SARS-CoV-2 outbreak in immune-mediated inflammatory diseases: the Euro-COVIMID multicentre cross-sectional study. Lancet Rheumatol. 2021 Jul;3(7):e481-e488. doi: 10.1016/S2665-9913(21)00112-0. Epub 2021 Apr 28. PMID 33942031